CLINICAL TRIAL: NCT00115050
Title: Open-label Safety Study of TMC114 in Combination With Low Dose RTV and Other ARVs in Highly Experienced HIV-1 Infected Patients With Limited or no Treatment Options.
Brief Title: TMC114-C209: A Study of Safety of TMC114 With Low Dose Ritonavir (RTV) and Other Antiretrovirals in Experienced HIV-1 Infected Patients With Limited or no Treatment Options
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002755
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV infections; Antiretroviral; TMC114; Ritonavir; Safety, TMC114-C209
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

INTERVENTIONS:
Drug: TMC114

SUMMARY:
This is an open-label safety study to provide early access to TMC114 for HIV-1 infected patients who have failed and exhausted regimens based on commercially available antiretroviral (ARV) therapy and who are ineligible for participation in any other Tibotec-sponsored trial.

DETAILED DESCRIPTION:
This is an open-label non-randomized safety study to provide early access to TMC114 for HIV-1 infected patients who have failed and exhausted regimens based on commercially available antiretroviral (ARV) therapy and who are ineligible for participation in any other Tibotec-sponsored trial. The safety and tolerability of TMC114 in combination with low dose ritonavir (RTV) and other ARVs in highly ARV-experienced HIV-1 infected patients with limited or no treatment options will be assessed. Treatment will be continued until treatment-limiting toxicity, lost to follow-up, withdrawal, pregnancy, discontinuation of TMC114 development or when TMC114 is commercially available to the patient. Total daily dose is 600 mg TMC114 twice daily, each intake in combination with one capsule of 100 mg Ritonavir. Since TMC114 is formulated as 300mg tablets (F014) this means 2X2 tablets per day, taken orally. Treatment will be continued until treatment-limiting toxicity, lost to follow-up, withdrawal, pregnancy, discontinuation of TMC114 development or when TMC114 is commercially available to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient has voluntarily signed the informed consent before initiation of study procedures
* Patient with documented HIV-1 infection
* Patient has limited or no treatment options because of multiple treatment failures
* Negative pregnancy test for females of childbearing potential
* CD4 cell count < or = 100 cells/mm³
* Viral load > or = 10,000 copies/mL.

Exclusion Criteria:

* Primary HIV infection, patient is eligible for other Tibotec-sponsored trials
* Prior or current participation in a trial with TMC114 (except for Phase I studies conducted in HIV-infected patients)
* Use of disallowed concomitant therapy
* Use of investigational medication during the trial or within the last 90 days
* Female patients who are pregnant or breast feeding or of child bearing potential without the use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last trial-related activity
* Patients with previously demonstrated clinically significant allergy or hypersensitivity to any or the excipients of the investigational medication (TMC114)
* Patients with the laboratory abnormalities as defined by a standardized grading scheme based on the Division of AIDS (DAIDS) table (updated version from December 2004) Any grade 3 or 4 toxicity with the following exceptions: Patients with pre-existing diabetes or asymptomatic glucose elevations of grade 3 or 4
* Patients with asymptomatic triglyceride elevations of grade 3 or 4, patients with clinical or laboratory evidence of active liver disease, liver impairment/dysfunction or cirrhosis irrespective or liver enzyme levels
* Note: Patients co-infected with chronic hepatitis B or C will be allowed to enter the trial if their condition is clinically stable. Patients diagnosed with acute viral hepatitis at screening will not be allowed to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to provide early access to TMC114 for highly ARV-experienced HIV-1 infected patients who have failed and exhausted treatment options based on commercially available ARVs

SECONDARY OUTCOMES:
The secondary objective is to gather additional information on the safety and tolerability of TMC114 in combination with low dose RTV and other ARVs.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Clinical Study Report Synopsis of TMC114-C209: A study of safety of TMC114 With Low Dose Ritonavir (RTV) and Other Antiretrovirals in Experienced HIV-1 Infected Patients With Limited or no Treatment Options — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=985&filename=CR002755_CSR.pdf